CLINICAL TRIAL: NCT03608774
Title: A Phase 4, Randomized, Double-Blinded, Placebo-Controlled Trial of Azithromycin Versus Doxycycline for the Treatment of Rectal Chlamydia in Men Who Have Sex With Men
Brief Title: Trial of Azithromycin vs. Doxycycline for the Treatment of Rectal Chlamydia in MSM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0092
Record Dates: First submitted 2018-06-28; First posted 2018-08-01 (Actual); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2019-01-25

CONDITIONS: Anal Chlamydia Infection
Keywords: Azithromycin; Doxycycline; Efficacy; MSM; Phase 4; Rectal Chlamydia
MeSH Terms: interventions — Azithromycin; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): 1 gram of Azithromycin (4 capsules of 250 mg) administered orally as a single dose on Day 1, and Doxycycline placebo (1 capsule) administered orally twice daily for 7 days starting on Day 1. N=123
  Interventions: Drug: Azithromycin; Other: Placebo
- Arm 2 (Experimental): 100 mg of Doxycycline (1 capsule) administered orally twice daily for 7 days starting on Day 1, and Azithromycin placebo (4 capsules) administered orally as a single dose on Day 1. N=123
  Interventions: Drug: Doxycycline; Other: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin monohydrate is a macrolide antibacterial drug, FDA-approved in the US for the treatment of Chlamydia trachomatis (CT) in dose 1 gram (4 capsules of 250 mg), administered orally as a single dose.
  Arms: Arm 1
Drug: Doxycycline — Doxycycline hyclate is an antibacterial drug synthetically derived from oxytetracycline, FDA-approved in the US for the treatment of Chlamydia trachomatis (CT) as a course of 100 mg (1 capsule), administered orally twice daily for 7 days.
  Arms: Arm 2
Other: Placebo — Azithromycin placebo (4 capsules), administered orally as a single dose; Doxycycline placebo (1 capsule), administered orally twice daily for 7 days.

SUMMARY:
A clinical trial to compare the efficacy of azithromycin (Arm 1) vs. doxycycline (Arm 2) administered per CDC's STD Treatment Guidelines for rectal Chlamydia trachomatis (CT) in men who have sex with men (MSM). Subjects will be males aged = / > 18 years with a microbiologically confirmed diagnosis of rectal CT and at least one male sex partner in the past 12 months. The trial will be conducted at two sites in the US and will enroll up to 274 total subjects to achieve 246 subjects who contribute to the primary analysis. The duration of this study will be approximately 16 months 22 months with subject participation duration 29 days. The primary objective of this study is to compare the efficacy of azithromycin vs. doxycycline for treatment of rectal CT infection in MSM based on microbiologic cure (negative NAAT) at Day 29.

DETAILED DESCRIPTION:
A Phase 4, multi-center, randomized, double-blinded, placebo-controlled trial to compare the efficacy of azithromycin (Arm 1) vs. doxycycline (Arm 2) administered per CDC's STD Treatment Guidelines for rectal Chlamydia trachomatis (CT) in men who have sex with men (MSM). The effect of Lymphogranuloma Venereum (LGV) infection on microbiologic cure in MSM with rectal CT will also be assessed. Arm 1 will comprise of subjects receiving 1 gram of Azithromycin (4 capsules of 250 mg) orally as a single dose, and Doxycycline placebo (1 capsule) orally twice daily for 7 days. Arm 2 will comprise of subjects receiving 100 mg of Doxycycline (1 capsule) administered orally twice daily for 7 days, and Azithromycin placebo (4 capsules) administered orally as a single dose. Subjects will be males aged = / >18 years with a microbiologically confirmed diagnosis of rectal CT and at least one male sex partner in the past 12 months. The trial will be conducted at two sites in the US and will enroll up to 274 total subjects to achieve 246 subjects who contribute to the primary analysis. The duration of this study will be approximately 22 months with subject participation duration 29 days. The primary objective of this study is to compare the efficacy of azithromycin vs. doxycycline for treatment of rectal CT infection in MSM based on microbiologic cure (negative NAAT) at Day 29. The secondary objectives are: 1) to assess the effect of LGV infection on microbiologic cure in MSM with rectal CT at Days 15 and 29 and 2) to compare the efficacy of azithromycin vs. doxycycline for treatment of rectal CT in MSM based on microbiologic cure at Day 15.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to understand and provide written informed consent before initiation of any study procedures.
2. Willing and able to comply with planned study procedures for all study visits.
3. Male sex at birth and aged = / > 18 years with valid contact information.
4. At least one male sex partner (oral or anal) in the past 12 months.
5. Untreated rectal CT diagnosed by a positive NAAT result.
6. Willingness to abstain from condomless receptive anal sex during the trial.
7. Willingness to complete a 7-day study drug regimen.

Exclusion Criteria:

1. Current clinical diagnosis of acute proctitis per the CDC's 2015 STD Treatment Guidelines: symptoms of anorectal pain, tenesmus, and/or rectal discharge with anoscopy findings confirming inflammation.
2. Concomitant untreated gonorrhea (rectal, pharyngeal, or urethral) or known exposure to gonorrhea in the time between CT testing and study enrollment.
3. Clinical diagnosis of concomitant untreated primary or secondary syphilis.
4. Known allergy to tetracyclines or macrolides.
5. Received antimicrobial therapy active against C. trachomatis within 21 days of positive rectal CT NAAT result, or between the positive CT NAAT result and study enrollment*.

   *This includes subjects treated empirically on the day of testing due to known exposure to gonorrhea or chlamydia, as well as enrollment in another study using antimicrobial therapy active against C. trachomatis, or planned enrollment in such a study during their time in this trial. Specifically, use of the following antibiotics is an exclusion criterion: azithromycin and other macrolides, doxycycline and related tetra- or glycylcyclines, fluoroquinolones, rifampin, quinupristin-dalfopristin, and linezolid.
6. Plans to move to another location that would preclude study follow-up appointments in clinic or by mail-in in the next 30 days.
7. Use of any investigational drug contraindicated to treatment with azithromycin or doxycycline within 7 days before enrollment.
8. Previous enrollment in this trial.
9. Any other condition that, in the opinion of the investigator, would interfere with participation in the trial.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fenway Health - The Fenway Institute, Boston, Massachusetts
  - University of Washington - Harborview Medical Center - Center for AIDS and STD, Seattle, Washington

REFERENCES:
- [Derived] Dombrowski JC, Wierzbicki MR, Newman LM, Powell JA, Miller A, Dithmer D, Soge OO, Mayer KH. Doxycycline Versus Azithromycin for the Treatment of Rectal Chlamydia in Men Who Have Sex With Men: A Randomized Controlled Trial. Clin Infect Dis. 2021 Sep 7;73(5):824-831. doi: 10.1093/cid/ciab153. PMID 33606009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for the study were men who have sex with men diagnosed with rectal chlamydia based on a positive rectal Chlamydia trachomatis (CT) nucleic acid amplification test (NAAT) result. The first participant was enrolled on 13 July 2018, and the last participant was enrolled in January 2020.
Groups:
- Azithromycin + Doxycycline Placebo: 1 gram of Azithromycin (4 capsules of 250 mg) administered orally as a single dose on Day 1, and Doxycycline placebo (1 capsule) administered orally twice daily for 7 days starting on Day 1. N=89
  Azithromycin: Azithromycin monohydrate is a macrolide antibacterial drug, FDA-approved in the US for the treatment of Chlamydia trachomatis (CT) in dose 1 gram (4 capsules of 250 mg), administered orally as a single dose.
  Placebo: Doxycycline placebo (1 capsule), administered orally twice daily for 7 days.
- Doxycycline + Azithromycin Placebo: 100 mg of Doxycycline (1 capsule) administered orally twice daily for 7 days starting on Day 1, and Azithromycin placebo (4 capsules) administered orally as a single dose on Day 1. N=88
  Doxycycline: Doxycycline hyclate is an antibacterial drug synthetically derived from oxytetracycline, FDA-approved in the US for the treatment of Chlamydia trachomatis (CT) as a course of 100 mg (1 capsule), administered orally twice daily for 7 days.
  Placebo: Azithromycin placebo (4 capsules), administered orally as a single dose.
Period: Overall Study
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Started | 89 | 88
Completed | 82 | 81
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Not eligible at enrollment | 0 | 1
Not completed — Health related event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized subjects, receiving or not receiving the study product, are included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (10.8) | 33.9 (11.6) | 33.7 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 89 | 88 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 21 | 37
  Not Hispanic or Latino | 71 | 67 | 138
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 10 | 12 | 22
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 3 | 5 | 8
  White | 54 | 58 | 112
  More than one race | 16 | 6 | 22
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 89 | 88 | 177
Rectal CT Symptomatic Status [Count of Participants; unit: Participants]
  Symptomatic | 18 | 13 | 31
  Asymptomatic | 71 | 74 | 145
  Not Available | 0 | 1 | 1
Inguinal Lymphadenopathy [Count of Participants; unit: Participants]
  Yes | 3 | 4 | 7
  No | 86 | 83 | 169
  Not Available | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) at Day 29
Description: Microbiologic cure was based on rectal CT (Chlamydia trachomatis) NAAT (nucleic acid amplification test) result. The proportion of subjects with microbiologic cure in each study arm at Day 29 is reported in this outcome measure.
Time Frame: Day 29
Population: The Complete Case population included randomized subjects who met all inclusion/exclusion criteria at enrollment, had a positive baseline rectal CT NAAT result, and had a Day 29 microbiologic result available.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 65 | 70
proportion of participants | 0.74 [0.56 to 0.86] | 1.00 [0.90 to 1.00]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Superiority; p < 0.001, Chi-squared — Protocol pre-specified an interim analysis of the primary outcome using O'Brien-Fleming bounds to maintain an overall 5% alpha level. The trial was stopped at the interim analysis. P-value was derived using stage-wise ordering of the sample space; Risk Difference (RD) = 0.26, 95% CI 2-sided [0.16 to 0.36] — Protocol pre-specified an interim analysis of the primary outcome using O'Brien-Fleming bounds to maintain an overall 5% alpha level. The trial was stopped at the interim analysis. Estimates were derived using stage-wise ordering of the sample space

2. Secondary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) at Day 15
Description: Microbiologic cure was based on rectal CT (Chlamydia trachomatis) NAAT (nucleic acid amplification test) result. The proportion of subjects with microbiologic cure in each study arm at Day 15 is reported in this outcome measure.
Time Frame: Day 15
Population: The Complete Case population included randomized subjects who met all inclusion/exclusion criteria at enrollment, had a positive baseline rectal CT NAAT result, and had a Day 15 microbiologic result available.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 67 | 70
proportion of participants | 0.84 [0.73 to 0.91] | 0.94 [0.86 to 0.98]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Other; Risk Difference (RD) = 0.11, 95% CI 2-sided [0.00 to 0.22]

3. Secondary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) Within the Subgroup of Non-LGV (Lymphogranuloma Venereum) Infected at Baseline
Description: Microbiologic cure was based on rectal CT (Chlamydia trachomatis) NAAT (nucleic acid amplification test) result. The proportion of subjects with microbiologic cure in each study arm at Day 15 is reported in this outcome measure. LGV strains of CT were identified via multiplex PCR (Polymerase Chain Reaction) on positive CT NAAT specimens.
Time Frame: Day 15
Population: The Complete Case population included randomized subjects who met all inclusion/exclusion criteria at enrollment, had a positive baseline rectal CT NAAT result, had a baseline LGV infection status result, and had a post-baseline microbiologic result available. Furthermore, participants in this subgroup analyses were non-LGV infected at baseline.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 63 | 66
proportion of participants | 0.84 [0.73 to 0.91] | 0.94 [0.85 to 0.98]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Other; Risk Difference (RD) = 0.10, 95% CI 2-sided [-0.01 to 0.21]

4. Secondary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) Within the Subgroup of Non-LGV (Lymphogranuloma Venereum) Infected at Baseline
Description: Microbiologic cure was based on rectal CT (Chlamydia trachomatis) NAAT (nucleic acid amplification test) result. The proportion of subjects with microbiologic cure in each study arm at Day 29 is reported in this outcome measure. LGV strains of CT were identified via multiplex PCR (Polymerase Chain Reaction) on positive CT NAAT specimens.
Time Frame: Day 29
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 61 | 66
proportion of participants | 0.74 [0.62 to 0.83] | 1.00 [0.94 to 1.00]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Other; Risk Difference (RD) = 0.26, 95% CI 2-sided [0.15 to 0.38]

5. Secondary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) Within the Subgroup of LGV (Lymphogranuloma Venereum) Infected at Baseline
Description: as for outcome 3
Time Frame: Day 15
Population: The Complete Case population included randomized subjects who met all inclusion/exclusion criteria at enrollment, had a positive baseline rectal CT NAAT result, had a baseline LGV infection status result, and had a post-baseline microbiologic result available. Furthermore, participants in this subgroup analyses were LGV infected at baseline.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 4 | 4
proportion of participants | 0.75 [0.30 to 0.95] | 1.00 [0.51 to 1.00]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Other; Risk Difference (RD) = 0.25, 95% CI 2-sided [-0.28 to 0.70]

6. Secondary Outcome: The Proportion of Subjects With Microbiologic Cure (Negative Rectal CT NAAT Result) Within the Subgroup of LGV (Lymphogranuloma Venereum) Infected at Baseline
Description: as for outcome 4
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
Number analyzed (Participants) | 4 | 4
proportion of participants | 0.75 [0.30 to 0.95] | 1.00 [0.51 to 1.00]
Statistical Analysis 1: Comparison: Azithromycin + Doxycycline Placebo vs Doxycycline + Azithromycin Placebo; Test type: Other; Risk Difference (RD) = 0.25, 95% CI 2-sided [-0.28 to 0.70]

ADVERSE EVENTS:
Time Frame: SAEs that occurred during the subject's participation in the trial (Day 1 through Day 29) were collected.
Description: Due to the safety profile of both drugs used in this trial, only SAEs (not non-serious AEs) that occurred after the first dose of treatment through Visit 3 (target at Day 29, visit window Day 25-31) were collected. SAEs included any untoward medical occurrence that resulted in death; was life threatening; required inpatient hospitalization or prolongation; or was a persistent/significant disability/incapacity. Participants considered at risk were restricted to those who received study product.
Arm/Group | Azithromycin + Doxycycline Placebo | Doxycycline + Azithromycin Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/87
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin + Doxycycline Placebo (N=89) | Doxycycline + Azithromycin Placebo (N=87)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT03608774/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03608774/SAP_001.pdf